CLINICAL TRIAL: NCT07027631
Title: Comparative Efficacy of Magnesium Sulfate Iontophoresis and Extracorporeal Shockwave Therapy on Chronic Mechanical Neck Pain. A Randomized Controlled Trial
Brief Title: Comparative Efficacy of Magnesium Sulfate Iontophoresis and Extracorporeal Shockwave Therapy on Chronic Mechanical Neck Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Al-Amir Mohamed Hussein, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeniSuefU24
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Mechanical Neck Pain
Keywords: shock wave therapy; Magnesium Sulfate iontophoresis; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium Sulfate Iontophoresis group (Experimental): Patients in this group will receive Magnesium Sulfate Iontophoresis, two sessions per week for four weeks
  Interventions: Device: Magnesium Sulfate Iontophoresis
- Shock Wave Therapy group (Experimental): Patients in this group will receive Shock Wave Therapy, one session per week for four weeks
  Interventions: Device: Shock Wave Therapy
- Control group (Placebo Comparator): Patients in this group will receive stretching and strengthening exercises, two sessions per week for four weeks
  Interventions: Other: stretching and strengthening

INTERVENTIONS:
Device: Magnesium Sulfate Iontophoresis — Magnesium Sulfate iontophoresis utilizing an iontophoretic drug delivery system
  Arms: Magnesium Sulfate Iontophoresis group
Device: Shock Wave Therapy — using Shock Wave Therapy Device
  Arms: Shock Wave Therapy group
Other: stretching and strengthening — stretching and strengthening exercises
  Arms: Control group

SUMMARY:
The purpose of the study is to investigate the Comparative Efficacy of Magnesium Sulfate Iontophoresis and Extracorporeal shockwave therapy on Chronic Mechanical Neck Pain

ELIGIBILITY:
Inclusion Criteria:

* medically competent men and women will be included
* They had chronic MTrPs in the upper trapezius for more than 6 months
* Diagnostic criteria of being a tight band with a palpable nodule and distant pain when subjected to pressure

Exclusion Criteria:

* subjects with previous neck or shoulder pathology (e.g., fracture, sur¬gery, inflammatory and infectious diseases),
* cervical disc pathology, systemic disorder, fibromyalgia,
* those who underwent physical therapy for at least the previous 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
pain pressure threshold | 0-4 weeks
  pain pressure threshold will be measured by the pressure algometer
Pain intensity | 0-4 weeks
  pain intensity will be measured by visual analogue scale

SECONDARY OUTCOMES:
Neck Disability Index | 0-4 Weeks
  Neck Disability Index is a questionnaire to measure function

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt